CLINICAL TRIAL: NCT06077448
Title: Role of Volumetric MRI Brain in Evaluation of Migraine
Brief Title: Volumetric MRI Brain in Patients With Migraine
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ann Basem Fathy Kamel, resident doctor, Assiut University
Other Study IDs: MRI brain in migraine
Record Dates: First submitted 2023-10-05; First posted 2023-10-11 (Actual); Last update posted 2023-10-11 (Actual); Status verified 2023-10

CONDITIONS: Migraine
MeSH Terms: conditions — Migraine Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- cases: patients with migraine (migraineurs)
  Interventions: Device: MRI
- controls: healthy individuals
  Interventions: Device: MRI

INTERVENTIONS:
Device: MRI — imaging modality

SUMMARY:
Assessment of the role of volumetric MRI in evaluation of different types of migraine .

DETAILED DESCRIPTION:
Migraine is a common condition that many people experience during their lives. Evolving data reported that migraine patients have increased risk of developing silent brain lesions, such as white matter lesions and volumetric changes in both grey and white matter found on MRI .

These changes have been first investigated with CT scans which reported cerebral edema, atrophy and ischemia . With the advent of MRI and high-resolution devices, the most commonly reported structural changes were white matter lesions .

Volumetric brain MRI is the tool segments and measures volumes of the key brain structures-hippocampus, ventricles and other structures-and compares the volumes to standard normal values based on age, gender and cranial volume. This information helps assess neurological conditions and neurodegenerative diseases .

* In migraine patients ,Volumetric MRI techniques allow better assessment of WMLs and may provide a different comprehension of structural aspects related to the migraine pathophysiology. The identification of migraineurs' brain structural alterations through non-invasive neuroimaging methods and the use of accessible and easy to-use software brings new perspectives on the assessment of the impact of this condition in central nervous system macro-architecture .
* In previous studies, structural brain changes in migraineurs were assessed by an automated segmentation using (Free Surfer) method .

In our study, we aim to investigate these total and segmental structural changes of brain volume in migraine patients; as well as white matter lesions, in comparison to healthy controls, and in patients with episodic migraine in comparison to chronic type of migraine using another automated tissue segmentation (Vol brain) method.

ELIGIBILITY:
Inclusion Criteria:

* Patients with different types of migraine :

  * episodic migraine without aura (MoA)
  * episodic migraine with aura (MA)
  * chronic migraine (CM).

Exclusion Criteria:

* . History of acute myocardial infarction, ischemic or hemorrhagic stroke. . History of neurosurgery or brain trauma

  * Patients with contra-indications to MRI.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The study will include migraine patients who visit headache out-patient clinic at Neuro-psychaitry Department Assuit University Hospital along 1 year compared to healthy controls.
Sampling Method: Non-Probability Sample
Enrollment: 66 (Estimated)
Dates: Start 2023-10-10 (Estimated); Primary Completion 2024-10-10 (Estimated); Study Completion 2025-02-01 (Estimated)

PRIMARY OUTCOMES:
To evaluate the role of volumetric MRI images in different types of migraine. | within first year of research
  to stand out accuracy of MRI to detect volumetric changes which affect brain tissue in migraine